CLINICAL TRIAL: NCT00411151
Title: An Open-label, Multicenter Phase II Trial of Sunitinib for Patients With Chemo-refractory Metastatic Gastric Cancer
Brief Title: Efficacy and Safety of Sunitinib in Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Markus Moehler, MD, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-SU-2006; KKS 2005-015
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2011-01-14 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Gastric Adenocarcinoma; Barrett Esophagus
Keywords: Adenocarcinoma of esophagogastric junction; Adenocarcinoma of lower esophagus (Barrett carcinoma)
MeSH Terms: conditions — Barrett Esophagus | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sunitinib-Malate — Capsules of 50, 25 or 12,5 mg. Dosage 50 mg, 37.5 mg or 25 mg once daily until progression of disease or untolerable side effects

SUMMARY:
This trial will be conducted to evaluate the efficacy, safety, and tolerability of sunitinib (sunitinib-malate) as a second-line palliative therapy in metastatic gastric cancer. Despite the efforts in front-line therapy, second-line protocols have not yet been established in randomized clinical trials for those patients. Although many patients are still in good performance status and present with low tumor burden after failure of first-line chemotherapy, they may clearly benefit from second-line treatment. Increasingly more metachronic metastatic patients are urging for new platinum-free therapeutic options due to the fast-growing use of (neo-) adjuvant platin-based protocols.

So far, only sparse data on chemotherapy are available after failure of platin-based protocols. Nearly only irinotecan-containing combinations have properly been analyzed, and produced excellent response rates and survival times of up to 30% and 7.6 months, respectively. However, irinotecan has not been approved yet for this indication. In addition, as irinotecan-containing regimens have been submitted for approval for first-line therapy, second-line regimens in irinotecan-refractory patients have not been evaluated in any trial. Thus, there is an urgent need to establish new second-line treatment options for both, cisplatinum- or irinotecan-combination refractory patients with advanced or metastatic gastric cancer.

Sunitinib inhibits the receptor tyrosine kinases (RTKs) involved in tumor proliferation and angiogenesis, specifically the VEGFR, PDGFR, KIT, FLT-3, and RET. The VEGF pathway has been shown to be a significant factor in metastatic gastric cancer. In gastric carcinoma cells, VEGF ligands and its receptors are definitely involved in the process of tumor progression. KDR and FLT-1 are expressed widely and VEGF stimulated KDR-positive tumor cell growth directly. The ligand VEGF-C has also been shown to be involved in progression of human gastric carcinoma, particularly via lymphangiogenesis. In addition, peritoneal metastases of some cancers such as gastric cancers were largely dependent on VEGF. Therefore, patients with chemo-refractory metastatic gastric cancer might benefit from VEGFR inhibitory therapy with sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent of the patient before the start of specific protocol procedures
* Histologically proven adenocarcinoma of stomach, esophagogastric junction or lower esophagus (Barrett carcinoma)
* Measurable metastatic disease according to the Response Evaluation Criteria in Solid Tumors (RECIST). If locally recurrent disease, it must be associated with at least one measurable lymph node (> 20 mm by computed tomography [CT] scan or > 10 mm with spiral CT).
* Failure of prior palliative chemotherapy/chemotherapies (at least one irinotecan- or cisplatin-based). Failure is defined either by progression of disease or by significant toxicity that precludes further treatment.
* At least 3 weeks from previous chemotherapy at first dose of trial drug
* Resolution of all acute toxic side effects of prior therapy or surgical procedures to grade ≤ 1 National Cancer Institute-Common Toxicity Criteria (NCI-CTC) (except for the laboratory values)
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin ≤ 1.5 x ULN
  * Absolute neutrophil count (ANC) ≥1500/microL
  * Platelets ≥ 100,000/microL
  * Hemoglobin ≥ 8.0 g/dL without support of growth factors (previous administration of erythrocyte concentrate is allowed)
  * Serum calcium ≤ 12.0 mg/dL
  * Serum creatinine ≤ 2.0 x ULN
  * Lipase/amylase ≤ 2.5 x ULN
  * All other laboratory values specified in the protocol (white blood cell count, white blood cell differential, alkaline phosphatase, sodium, potassium, creatinine clearance): resolution of all side effects of prior therapy or surgical procedure to grade < 3 NCI-CTC
* At least 4 weeks from any major surgery (at first dose of trial drug)
* Karnofsky Performance Status (KPS) ≥ 70
* Life expectancy > 12 weeks
* Patients must be able to swallow sunitinib capsules
* Patients who understand the nature of the trial and are willing and able to comply with scheduled visits, treatment plans, laboratory tests and other trial procedures
* Female patients who are capable of bearing children must have a negative pregnancy test result (serum or urine) at trial entry. All women included in the trial must be surgically sterile or postmenopausal or agree to employ adequate birth control measures for the duration of the trial and six months post-dosing. Male patients must be surgically sterile or must agree to use effective contraception during the trial and six months post-dosing.

Exclusion Criteria:

* Tumor type other than adenocarcinoma (e.g., leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix which has been effectively treated. Patients curatively treated and disease free for at least 5 years will be discussed with the sponsor before inclusion.
* Patients with known brain or leptomeningeal metastasis
* Intake of non-permitted concomitant drugs. (The coordinating investigator should be contacted to discuss the individual case.)

  * Concomitant treatment with antiarrhythmics and drugs with dysrhythmic potential (i.e., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, and indapamide)
  * Administration of potent CYP34A inhibitors during or within 7 days before start of sunitinib-treatment (e.g. ketoconazole, itraconazole, clarithromycin, erythromycin, diltiazem, verapamil, delavirdine, indinavir, saquinavir, ritonavir, atazanavir, nelfinavir, grapefruit juice)
  * Administration of potent CYP3A4 inducers during or within 12 days before start of sunitinib-treatment (e.g. dexamethasone, rifampicin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John´s wort, efavirenz, tipranavir)
  * Ongoing treatment with therapeutic doses of anticoagulants such as Coumadin or heparins. (However, low dose Coumadin up to 2 mg by mouth [PO] daily for deep vein thrombosis prophylaxis is allowed.)
  * Any other medicinal anticancer therapy during treatment phase except treatment with non-conventional therapies (e.g. herbs or acupuncture) and vitamins/mineral supplements, provided that they do not interfere with the trial endpoint, in the opinion of the investigator
  * Concurrent systemic immune therapy, chemo- or hormone therapy
  * Concomitant or within a 4-week period administration (from first dose of trial drug) of any other experimental drug under investigation (except for irinotecan and cetuximab) and participation in another clinical trial
* Any prior radiotherapy of target lesions
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (> hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis
* Current history of chronic diarrhoea
* Active disseminated intravascular coagulation, or patients prone to thromboembolism
* Any of the following events (in any grade) prior to starting the trial treatment:

  * myocardial infarction
  * severe/unstable angina
  * coronary/peripheral artery bypass graft
  * congestive heart failure
  * cerebrovascular accident or transient ischemic attack
  * pulmonary embolism
* Known history of QT interval prolongation, ongoing QT prolongation (> 450 msec for males or > 470 msec for females), any cardiac ventricular dysrhythmias, atrial fibrillation of any grade
* Hypertension that cannot be controlled by medications (> 150/100 mmHg despite optimal medical therapy)
* Known human immunodeficiency virus (HIV) infection
* Active uncontrolled infection
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with trial participation or trial drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into the trial
* Pregnant or lactating women
* Known allergic/hypersensitivity reaction to any of the components of the treatment; or known drug abuse/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, MD, Principal Investigator — Johannes-Gutenberg-University of Mainz, I. Dept. Internal Medicine
Locations (12):
- Germany (12):
  - Universität Heidelberg, Nationales Zentrum für Tumorerkrankungen, Heidelberg, Baden-Würtemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Würtemberg
  - TU München, Klinikum rechts der Isar, II. Med. Klinik und Poliklinik, München, Bavaria
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Universitätsklinik zu Köln, Klinik I für Innere Medizin, Cologne, North Rhine-Westphalia
  - Universitätsklinikum der GHS Essen, Innere Klinik und Poliklinik, Tumorforschung, Essen, North Rhine-Westphalia
  - Klinikum der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland
  - Universitätsklinikum Carl Gustav Carus, Med. Klinik I, Dresden, Saxony
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité, Campus Benjamin Franklin, Berlin, State of Berlin
  - KH Nordwest, Abteilung für Hämatologie und Onkologie, Frankfurt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in (FPI): 15.02.2007 Last patient out (LPO): 20.08.2009
Groups:
- Sunitinib: open-label and uncontrolled treatment cycle "4+2": Sunitinib capsules for oral administration (50mg daily for 4 weeks and 2 weeks rest)
Period: Overall Study
Arm/Group | Sunitinib
Started | 52
Completed | 5
Not Completed | 47
Not completed — Death | 38
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Trial prematurely closed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 52
Age Continuous [Median (Full Range); unit: years] | 59 (12.07) [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 40
Karnofsky Performance Status (KPS) [Number; unit: Participants] — KPS is the Karnofsky Lansky Score. Higher values in the KPS represent a better physical condition. 100%=normal, 90%=able to carry on normal activity, 80%=normal activity with effort, 70%=cares for self but unable to carry on normal activity, 60%=requires occasional assistance, 50%=requires considerable assistance and frequent medical care, 40%=disabled, requires special care and assistance, 30%=severely disabled and hospitalization indicated but death not imminent, 20%=very sick and requires hospitalization, 10%=moribund and fatal processes progressing rapidly, 0%=dead
  Participants
    100% | 17
    90% | 15
    80% | 18
    70% | 2
    60% | 0
    50% | 0
    40% | 0
    30% | 0
    20% | 0
    10% | 0
    Missing | 0
Localisation of adenocarcinoma [Number; unit: Participants] — Note that multiple answers are permitted.
  Participants
    Stomach | 36
    Gastroesophageal junction | 12
    Lower esophagus | 5
    Missing | 0
Grading of adenocarcinoma [Number; unit: Participants] — Grading of adenocarcinoma is the tumor grading according to UICC.
  1 (low grade)=well differentiated, 2 (intermediate grade)=differentiated, 3 (high grade)=poorly differentiated, 4 (high grade)=undifferentiated
  Participants
    1 | 0
    2 | 19
    3 | 26
    4 | 2
    Missing | 5
Localisation of target lesions [Number; unit: Participants] — Note that multiple answers are permitted.
  Participants
    Primary tumor | 3
    Lung | 8
    Liver | 28
    Lymph node truncus coeliacus | 10
    Lymph node mediastinum | 11
    Lymph node spleen/pancreas | 3
    Lymph node paraaortal caudal | 9
    Peritoneum | 2
    Soft tissue | 5
    Other | 14
    Missing | 0
Total size of target lesions [Median (Full Range); unit: mm] | 62 [10 to 236]
Localisation of non-target lesions [Number; unit: Participants] — Note that multiple answers are permitted.
  Participants
    Primary tumor | 1
    Bone | 1
    Lung | 4
    Liver | 15
    Lymph node truncus coeliacus | 4
    Lymph node mediastinum | 3
    Lymph node paraaortal caudal | 3
    Peritoneum | 3
    Other | 9
    No non-target lesions | 9
    Missing | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The primary endpoint is the ORR within the first 6 treatment cycles, defined as the percentage of participants with a confirmed reduction in tumor size fulfilling the criteria for complete or partial response (CR or PR) according to RECIST. CR=disappearance of all target lesions, PR=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions
Time Frame: one year
Population: Intention-to-treat (ITT) population comprises all patients registered, except one patient whose tumor diagnosis was not confirmed.
Measure: Number (95% Confidence Interval); unit: Participants (%)
Arm/Group | Sunitinib
Number analyzed (Participants) | 51
Participants (%) | 3.92 [0.48 to 13.46]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from first dose of trial medication to first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Time Frame: one year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 51
Days | 39 [36 to 58]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of trial medication to date of death due to any cause.
Time Frame: one year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sunitinib
Number analyzed (Participants) | 51
Days | 177 [106 to 278]

4. Secondary Outcome: One-Year Survival
Description: One-year survival is defined as the percentage of participants surviving for at least one year after first dose of trial medication.
Time Frame: one year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Participants (%)
Arm/Group | Sunitinib
Number analyzed (Participants) | 51
Participants (%) | 23.7 [12.8 to 36.5]

5. Secondary Outcome: Adverse Events
Description: The number of participants with at least one adverse event was measured.
Time Frame: one year
Population: Safety population comprises all patients registered.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 52
Participants | 52

6. Secondary Outcome: Safety and Tolerability: Serious Adverse Events
Description: The number of participants with at least one Serious Adverse Event was measured.
Time Frame: one year
Population: Safety population comprises all patients registered.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 52
Participants | 26

7. Secondary Outcome: Safety and Tolerability: Adverse Events in ≥10% of Patients
Time Frame: one year
Population: Safety population comprises all patients registered.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 52
Participants
  Fatigue | 19
  Nausea | 16
  Mucosal inflammation | 9
  Anorexia | 9
  Vomiting | 8
  Diarrhoea | 8
  Dysgeusia | 6
  Headache | 5
  Paraesthesia | 5
  Cough | 5
  Abdominal pain | 5
  Palmar-plantar erythrodysaesthesia syndrome | 5
  Blood bilirubin increased | 5
  Leukopenia | 11
  Thrombocytopenia | 11
  Neutropenia | 8
  Anaemia | 7

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes